CLINICAL TRIAL: NCT02646111
Title: An Open-label, Multi-center Study to Evaluate Sustained Virologic Response With Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir With and Without Ribavirin in Genotype 1 Chronic Hepatitis C Virus Infected Patients With Past PI Failure
Brief Title: Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir With and Without Ribavirin in Protease-Inhibitors ("PI") Failures
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Research and Development manager, Tel-Aviv Sourasky Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-15-OS-503-CTIL
Record Dates: First submitted 2015-12-28; First posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Hepatitis C
Keywords: "Hepatitis C Virus"; "Triple Therapy"; "PI Failure"; "Genotype 1"
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Genotype 1b without cirrhosis (Experimental): 12 weeks without Ribavirin
  Interventions: Drug: 12 weeks without Ribavirin
- Genotype 1b with cirrhosis (Experimental): 12 weeks with Ribavirin
  Interventions: Drug: 12 weeks with Ribavirin
- Genotype 1a without cirrhosis (Experimental): 12 weeks with Ribavirin
  Interventions: Drug: 12 weeks with Ribavirin
- Genotype 1a with cirrhosis (Experimental): 24 weeks with Ribavirin
  Interventions: Drug: 24 weeks with Ribavirin

INTERVENTIONS:
Drug: 12 weeks without Ribavirin — 12 weeks Triple Therapy: Ombitasvir, Paritaprevir, Ritonavir (25/150/100 mg dose) once daily and Dasabuvir 250 mg twice daily.
  Other Names: Triple therapy
  Arms: Genotype 1b without cirrhosis
Drug: 12 weeks with Ribavirin — 12 weeks Triple Therapy: Ombitasvir, Paritaprevir, Ritonavir 25/150/100 mg dose once daily + Dasabuvir 250 mg twice daily + weight adjusted Ribavirin, daily dose: 1,000 mg weight <75 kg, 1,200 mg weight> 75 kg.
  Other Names: Triple therapy
  Arms: Genotype 1a without cirrhosis; Genotype 1b with cirrhosis
Drug: 24 weeks with Ribavirin — 24 weeks Triple Therapy: Ombitasvir, Paritaprevir, Ritonavir 25/150/100 mg dose once daily + Dasabuvir 250 mg twice daily + weight adjusted Ribavirin, daily dose: 1,000 mg weight <75 kg, 1,200 mg weight> 75 kg.
  Other Names: Triple therapy
  Arms: Genotype 1a with cirrhosis

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of triple therapy of AbbVie adults with chronic hepatitis C virus ("HCV"), who have not responded to prior treatment with protease inhibitors.

The "Triple therapy" of AbbVie attacks various sites of the viral genome, thus increasing the potential efficacy of the treatment, especially for patients who have failed PI treatment.

DETAILED DESCRIPTION:
Patients with genotype 1 HCV, who underwent past triple therapy (Telaprevir, Boceprevir or Simeprevir with Pegylated interferon / Ribavirin) and are non-responders, partial responders or in relapse - will be screened in all research centers up to 30 days before the first treatment.

At the end of the initial assessment - the recruited participants will be allocated to different treatment groups in accordance with the hepatitis virus subtype 1a, 1b and presence of cirrhosis, as follows:

* Group A - genotype 1b without cirrhosis - 12 weeks of treatment *
* Group B - genotype 1b with cirrhosis - 12 weeks of treatment
* Group C - genotype 1a without cirrhosis - 12 weeks of treatment
* Group D - genotype 1a with cirrhosis - 24 weeks of treatment

(* Only this group will not get Ribavirin)

During the treatment period, participants will be asked to describe the treatment's tolerability (in terms of side effects) using self-administered questionnaires: SF-36, and WPAI Hep C v2.0.

The follow up will also include physical assessments, side effects documentation, blood tests, abdominal Ultrasound and Fibroscan.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hepatitis C, genotype 1A or 1B.
* Documentation of PI failure of treatment at least 12 months prior to study entry.
* Patients with cirrhosis - (only patients with cirrhosis Child A with only 5 points).

Exclusion Criteria:

* Inability to stay in the study for 36 weeks.
* Diagnosis of cross-contamination by HIV or Hepatitis B virus.
* Renal disfunction (creatinine clearance <30 ml / min).
* Evidence of hepatic carcinoma.
* Another serious disease, which may interfere with the study.
* Pregnant / breast-feeding women.
* Men with pregnant partners.
* Drug or alcohol abuse in the six months preceding the study.
* Chronic liver disease other than hepatitis C (such as Primary biliary cirrhosis, Primary sclerosing cholangitis, Autoimmune hepatitis).
* Current other treatment for HCV.
* Past PI Failure due to adverse events.
* Patients with cirrhosis Child B.
* Patients with cirrhosis, who were at child B and improved to child A after treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
"SVR" (sustained virologic response) rates | 12 weeks after end of treatment
  Sustained virologic response

SECONDARY OUTCOMES:
"SF" (short-form)-36 health survey | Day 1, weeks 4, 12, 24, 36.
  psychometrically-based physical and mental health and a preference-based health utility index.
WPAI Hep C v2.0 questionnaire | Day 1, weeks 4, 12, 24, 36.
  a scoring manual for work productivity and activity impairment assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Oren Shibolet, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Deutsch L, Houri I, Ben-Ari Z, Shlomai A, Veitsman E, Cohen-Ezra O, Issachar A, Mor O, Gozlan Y, Bruck R, Menachem Y, Zelber-Sagi S, Katchman H, Shibolet O. Ombitasvir/paritaprevir/ritonavir & dasabuvir +/- ribavirin following protease inhibitors failure - a prospective multi-centre trial. BMC Infect Dis. 2020 Apr 3;20(1):264. doi: 10.1186/s12879-020-4921-3. PMID 32245397